CLINICAL TRIAL: NCT04733989
Title: Development of a Biomarker Database to Investigate Aß, P-tau, and NfL Blood-Based Biomarkers and Digital Biomarkers in Older Participants Screened for Preclinical Alzheimer's Disease (AD), Prodromal AD, or Mild AD
Brief Title: A Biomarker Database to Investigate Blood-Based and Digital Biomarkers in Participants Screened for Alzheimer's Disease (Bio-Hermes)
Status: Completed | Type: Observational
Sponsor: GAP Innovations, PBC (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO-HERMES-001
Record Dates: First submitted 2020-12-28; First posted 2021-02-02 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease; Alzheimer Disease, Early Onset; Mild Cognitive Impairment; Memory Loss; Memory Disorders; Memory Impairment
Keywords: Alzheimer's disease; Alzheimer Disease, Early Onset; Mild Cognitive Impairment; Memory Loss; Memory Disorders; Memory Impairment; Older Volunteers; Healthy Volunteers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Beta-Amyloid, Phospho-Tau, Neurofilament Light Chain, DNA, RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarker Data Collection — During this study, a sample of your blood will be collected and you will have a PET scan taken of your brain. Blood sample results will be compared to PET scan pictures to understand how well the markers in the blood predict whether there is amyloid in the brain. Blood samples will also be collected that contain your genes. These genetic samples will also be compared to PET scans to help researchers understand how different people react to medicines and to understand the genetic causes of Alzheimer's disease. Some of the samples will be stored for future analysis.

SUMMARY:
The purpose of this study (Bio-Hermes) is to develop a blood, digital, and brain amyloid PET scan biomarker database that can be used to determine whether a meaningful relationship exists between digital tests, blood amyloid-beta, p-tau, and neurofilament biomarker levels and amyloid-beta levels identified through brain amyloid PET images. Blood collected will also be genetically sequenced to gain insights about genes and brain amyloid. The Bio-Hermes study will include 1,000 volunteers over the age of 60 screened for Preclinical Alzheimer's Disease, Prodromal AD, or Mild Dementia AD, and includes an endpoint enrollment requirement of 200 participants from underrepresented minority populations.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria for entry into the study:

1. Participants must provide written consent in the IRB-approved informed consent form or have a Legally Authorized Representative (LAR) provide written consent in the IRB-approved consent form on the participant's behalf;
2. Male or female 60 to 85 years of age (inclusive) at the time of consent;
3. Participants must be willing to undergo an amyloid PET scan within 60 days of signing informed consent; or for sites that do not have access to PET imaging, the participant must be willing to undergo a lumbar puncture for cerebrospinal fluid (CSF) collection within 30 days of the coagulation panel;
4. Participants must have a study partner who, in the investigator's judgement, has sufficient and frequent contact (defined as at least 8 hours of contact a week) with the participant and is able to provide accurate information regarding the participant's cognitive and functional abilities;
5. Participants must be willing to comply with all study procedures as outlined in the informed consent, including blood sampling;
6. Fluency in the language of the tests used at the study site;
7. Participants must be willing to be contacted for possible participation in clinical research trials once their participation in this study ends; and
8. Participants must have a Mini-Mental State Exam (MMSE) score of 17 to 30 inclusive at screening; those with a score of 17-19 must have a diagnosis of Probable AD.

Exclusion Criteria

Participants who meet any of the following criteria will not be eligible for entry into the study:

1. Participants who, in the opinion of the Site Principal Investigator, have serious or unstable medical conditions that would prohibit their completion of all study procedures and data collection;
2. Participants who have serious or unstable medical conditions that would likely preclude their participation in an interventional research trial;
3. Participants who are unable to undergo amyloid PET due to self-reported pregnancy, sensitivity of ligands being used, poor venous access, contraindication to PET, or planned or recent exposure to ionizing radiation that in combination with the planned administration of amyloid radioligand would result in a cumulative exposure that exceeds recommended local guidelines;
4. Participants who have reported or have a known negative amyloid PET scan in past 12 months;
5. Participants with self-reported, untreated conditions such as vitamin B12 or folate deficiency or bladder infections that in the opinion of the Site Principal Investigator could contribute to cognitive impairment;
6. Participants with history of stroke or seizures within 1 year of the Visit 1 (Screening);
7. Participants with history of cancer within the past 5 years with the exception of non-melanoma skin cancer or prostate cancer in situ;
8. Participants with known or suspected alcohol or drug abuse or dependence within 1 year of the Visit 1 (Screening);
9. Participants who report any current unstable psychiatric symptoms that could interfere with study procedures or impact study data (e.g., uncontrolled depression);
10. Participants who have participated in a clinical trial of any potential disease modifying AD treatment and received active drug within 6 months prior to Visit 1 (Screening);
11. Participants who have completed clinical or observational study procedures (e.g., imaging, cognitive testing) within 3 months of Visit 1 (Screening);
12. Participants who have any neurological disorder affecting the central nervous system, other than AD, that may be contributing to cognitive impairment (e.g., Parkinson's disease, other dementias, multiple concussions or seizures) as deemed significant by the Site Principal Investigator;
13. Participants with a Geriatric Depression Scale (GDS) score greater than or equal to 8 at Visit 1 (Screening);
14. Participants with a RAVLT-Delayed Recall Score of 1.5 standard deviation above the age-adjusted mean;
15. Participants with known history or self-report to be Human Immunodeficiency Virus (HIV) Positive;
16. Participants weighing less than 110 pounds;
17. Participants that have previously been consented to this study unless prior approval was granted by the Sponsor on a case-by-case basis;
18. Participants who are direct employees or family members of direct employees of the participating investigators' sites;
19. Participants who are direct employees of the Sponsor;
20. Participants who, in the opinion of the investigator, are unable to complete cognitive testing due to inadequate visual or auditory acuity;
21. For participants of the RetiSpec retinal substudy only: Those with a known history of ocular diseases (such as retinopathy, age-related macular degeneration, and glaucoma), with the exception of mild to moderate cataracts, and/or vision correction with glasses/contact lenses;
22. For participants undergoing LP: contraindication to lumbar puncture, including coagulopathy, concomitant anticoagulation (except for a platelet inhibitor such as aspirin or clopidogrel), thrombocytopenia, prior lumbar spinal surgery, significant deformity of the lumbosacral region, INR results > 1.3, or other factor that precludes safe LP in the opinion of the Site Principal Investigator.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1,000 participants
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Measurement of each participant's blood-based biomarker (Beta-Amyloid, Phospho-Tau, Neurofilament Light Chain) levels will be collected through blood sampling. | Through study completion, an average of 1 year
Measurement of each participant's amyloid levels in the brain will be collected through amyloid PET brain scan imaging. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Visionary Investigators Network - Aventura, Aventura, Florida
  - Visionary Investigators Network - Coral Gables, Coral Gables, Florida
  - Charter Research - Lady Lake, Lady Lake, Florida
  - JEM, Lake Worth, Florida
  - ClinCloud, Maitland, Florida
  - Visionary Investigators Network - South Miami, Miami, Florida
  - K2, Orlando, Florida
  - Visionary Investigators Network - Pembroke Pines, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Charter Research - Winter Park, Winter Park, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Kansas University Alzheimer's Disease Center (KUADC), Fairway, Kansas
  - Velocity Clinical Research - Syracuse, Syracuse, New York
  - Kerwin Research Center, Dallas, Texas
  - El Faro Health and Therapeutics, Rio Grande City, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baek MJ, Kim K, Park YH, Kim S. The Validity and Reliability of the Mini-Mental State Examination-2 for Detecting Mild Cognitive Impairment and Alzheimer's Disease in a Korean Population. PLoS One. 2016 Sep 26;11(9):e0163792. doi: 10.1371/journal.pone.0163792. eCollection 2016. PMID 27668883
- [Background] Berry CC. A tutorial on confidence intervals for proportions in diagnostic radiology. AJR Am J Roentgenol. 1990 Mar;154(3):477-80. doi: 10.2214/ajr.154.3.2106207. No abstract available.
- [Background] Cahn-Hidalgo D, Estes PW, Benabou R. Validity, reliability, and psychometric properties of a computerized, cognitive assessment test (Cognivue(R)). World J Psychiatry. 2020 Jan 19;10(1):1-11. doi: 10.5498/wjp.v10.i1.1. eCollection 2020 Jan 19. PMID 31956523
- [Background] Chetelat G, La Joie R, Villain N, Perrotin A, de La Sayette V, Eustache F, Vandenberghe R. Amyloid imaging in cognitively normal individuals, at-risk populations and preclinical Alzheimer's disease. Neuroimage Clin. 2013 Mar 5;2:356-65. doi: 10.1016/j.nicl.2013.02.006. eCollection 2013. PMID 24179789
- [Background] Giri M, Zhang M, Lu Y. Genes associated with Alzheimer's disease: an overview and current status. Clin Interv Aging. 2016 May 17;11:665-81. doi: 10.2147/CIA.S105769. eCollection 2016. PMID 27274215
- [Background] Howell JC, Watts KD, Parker MW, Wu J, Kollhoff A, Wingo TS, Dorbin CD, Qiu D, Hu WT. Race modifies the relationship between cognition and Alzheimer's disease cerebrospinal fluid biomarkers. Alzheimers Res Ther. 2017 Nov 2;9(1):88. doi: 10.1186/s13195-017-0315-1. PMID 29096697
- [Background] Ingelfinger, JA, Mosteller, R, Thibodeau, LA, Ware, JA. Biostatistics in Clinical Medicine. 3rd ed. New York, N.Y.: McGraw-Hill, New York; 1994.
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Kantarci K. Molecular imaging of Alzheimer disease pathology. AJNR Am J Neuroradiol. 2014 Jun;35(6 Suppl):S12-7. doi: 10.3174/ajnr.A3847. Epub 2014 Feb 6. PMID 24503555
- [Background] Malzbender K, Lavin-Mena L, Hughes L, Bose N, Goldman D, Patel D. White Paper on Key Barriers to Clinical Trials for Alzheimer's Disease. USC Schaeffer Center for Health Policy & Economics and Gates Ventures. August 2020. https://healthpolicy.usc.edu/wp-content/uploads/2020/08/Key-Barriers-to-Clinical-Trials-for-Alzheimer%E2%80%99s-Disease_FINAL.pdf. Accessed December 01, 2020.
- [Background] Morris JC, Schindler SE, McCue LM, Moulder KL, Benzinger TLS, Cruchaga C, Fagan AM, Grant E, Gordon BA, Holtzman DM, Xiong C. Assessment of Racial Disparities in Biomarkers for Alzheimer Disease. JAMA Neurol. 2019 Mar 1;76(3):264-273. doi: 10.1001/jamaneurol.2018.4249. PMID 30615028
- [Background] Niemantsverdriet E, Valckx S, Bjerke M, Engelborghs S. Alzheimer's disease CSF biomarkers: clinical indications and rational use. Acta Neurol Belg. 2017 Sep;117(3):591-602. doi: 10.1007/s13760-017-0816-5. Epub 2017 Jul 27. PMID 28752420
- [Background] O'Bryant SE, Humphreys JD, Smith GE, Ivnik RJ, Graff-Radford NR, Petersen RC, Lucas JA. Detecting dementia with the mini-mental state examination in highly educated individuals. Arch Neurol. 2008 Jul;65(7):963-7. doi: 10.1001/archneur.65.7.963. PMID 18625866
- [Background] US Food and Drug Administration. De Novo Classification Request For Cognivue. De Novo Summary (DEN130033). www.accessdata.fda.gov/cdrh_docs/reviews/DEN130033.pdf. Accessed December 7, 2020.
- [Background] Weiner MW, Veitch DP, Aisen PS, Beckett LA, Cairns NJ, Green RC, Harvey D, Jack CR Jr, Jagust W, Morris JC, Petersen RC, Saykin AJ, Shaw LM, Toga AW, Trojanowski JQ; Alzheimer's Disease Neuroimaging Initiative. Recent publications from the Alzheimer's Disease Neuroimaging Initiative: Reviewing progress toward improved AD clinical trials. Alzheimers Dement. 2017 Apr;13(4):e1-e85. doi: 10.1016/j.jalz.2016.11.007. Epub 2017 Mar 22. PMID 28342697
- [Background] Zhang J, Zhou W, Cassidy RM, Su H, Su Y, Zhang X; Alzheimer's Disease Neuroimaging Initiative. Risk factors for amyloid positivity in older people reporting significant memory concern. Compr Psychiatry. 2018 Jan;80:126-131. doi: 10.1016/j.comppsych.2017.09.015. Epub 2017 Oct 6. PMID 29091778
- [Derived] Galvin JE, Kleiman MJ, Harris HM, Estes PW. The Cognivue Amyloid Risk Measure (CARM): A Novel Method to Predict the Presence of Amyloid with Cognivue Clarity. Neurol Ther. 2025 Jun;14(3):865-880. doi: 10.1007/s40120-025-00741-x. Epub 2025 Apr 7. PMID 40192926
- [Derived] Galvin JE, Kleiman MJ, Estes PW, Harris HM, Fung E. Cognivue Clarity characterizes mild cognitive impairment and Alzheimer's disease in biomarker confirmed cohorts in the Bio-Hermes Study. Sci Rep. 2024 Oct 18;14(1):24519. doi: 10.1038/s41598-024-75304-5. PMID 39424626
- [Derived] Jannati A, Toro-Serey C, Gomes-Osman J, Banks R, Ciesla M, Showalter J, Bates D, Tobyne S, Pascual-Leone A. Digital Clock and Recall is superior to the Mini-Mental State Examination for the detection of mild cognitive impairment and mild dementia. Alzheimers Res Ther. 2024 Jan 2;16(1):2. doi: 10.1186/s13195-023-01367-7. PMID 38167251